CLINICAL TRIAL: NCT02965196
Title: Dexamethasone Therapy for Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HY-78-16
Record Dates: First submitted 2016-11-13; First posted 2016-11-16 (Estimated); Last update posted 2016-11-16 (Estimated); Status verified 2016-11

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexamethasone Therapy (Active Comparator): Three consecutive doses of IV Dexamethasone with be administered over three days. The doses will be tapered according to the following: 1st dose, 26mg., 2nd dose, 20mg., and the third dose will be 10 mg. Each dose will be administered over 24 hours in a slow drip, in a 100cc. normal saline bag (0.9%).
  Interventions: Drug: IV Dexamethasone Therapy
- Placebo Therapy (Placebo Comparator): Three consecutive doses of 100cc IV normal saline (0.9%), will be administered over three days. Each dose will be administered over 24 hours in a slow drip.
  Interventions: Other: IV Normal Saline (NaCl 0.9%)

INTERVENTIONS:
Drug: IV Dexamethasone Therapy
  Arms: Dexamethasone Therapy
Other: IV Normal Saline (NaCl 0.9%)
  Arms: Placebo Therapy

SUMMARY:
The study will evaluate the efficacy of IV Dexamethasone in treatment low back pain as an adjunct to analgesics.

ELIGIBILITY:
Inclusion Criteria:

* No "red flags" of serious spinal pathology
* Normal neurological examination
* Indication for opioid analgesia based on our pain management protocol
* No known hypersensitivity to the medication
* Ability to provide informed consent

Exclusion Criteria:

* Pregnancy
* All others who do not meet inclusion criteria

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Pain Reduction | Four days
  Pain will be measured according to the Visual Analog Scale throughout the treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel

IPD SHARING:
Plan to Share IPD: No